CLINICAL TRIAL: NCT02866318
Title: CUSUM Analysis in the Assessment of Novice Practitioners' Visual Estimation in LV Ejection Fraction With Echocardiographic Images
Brief Title: Learning Curve CUSUM of LV Ejection Fraction by Visual Estimation in Novice Practitioners
Acronym: LCCUSUMLVEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Fellowship, Emergency Medincine, Hanyang University
Other Study IDs: LCCUSUMchallenge1
Record Dates: First submitted 2016-03-08; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Novice practitioners: Residents in Emergency department who has no experiences of echocardiography prior to the study.
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography

SUMMARY:
This retrospective, cross-sectional cohort study was conducted to investigate the novice practitioners' learning curve of visual estimation of LV ejection fraction (%) through a echocardiographic video files at the academic emergency department (ED) in tertiary urban hospital.

DETAILED DESCRIPTION:
Eight EM residents who have no experience of echocardiography prior to the study were recruited as analysis of the echocardiographic image file. They received echocardiography interpretation skill training which included one hour of lecture. Twenty echocardiography videos files were provided during training session, they were instructed how to estimate EF by looking at the LV contractility without taking any measurement.

This procedure took less than 2 minutes in each case. An evaluation form was completed by each EP. EF is estimated qualitatively (Normal / Global hypokinesia), RWMA and quantitatively (%) by EP with echocardiographic certification(cardiologist). An each echocardiography has been performed with M7R® model ultrasound machine was reported by experienced echocardiographers as using MSM. The echocardiography results were reported blinded to our study.

A participant estimated the EF based on a complete assessment of LV wall motion including parasternal long-axis, short-axis, and apical four chamber view except for MSM.

And, participants wrote down EF(%) and a region of WMA as visual assessment and checked Normal wall motion or Global hypokinesia in EF reporting paper.

ELIGIBILITY:
Inclusion Criteria:

* EM residents who have no experience of echocardiography

Exclusion Criteria:

* They do not want to participate this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eight EM residents who have no experience of echocardiography prior to the study were recruited as analysis of the echocardiographic image file.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Learning curve | 2 hours
  Rate of concordance

CONTACTS AND LOCATIONS:
Overall Officials: YOONJE LEE, M.D., Principal Investigator — Hanyang University Guri Hospital
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes